CLINICAL TRIAL: NCT01844466
Title: Correlation of Visual and Motor Deficits in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Avraam Ploumis, Assistant Professor of PMR Surgical Dept, University of Ioannina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38/3-10-2011
Record Dates: First submitted 2013-04-24; First posted 2013-05-01 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Stroke
Keywords: course of motor and visual rehabilitation; improvement of deficits; stroke patients
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities; Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- stroke patients (Experimental)
  Interventions: Procedure: Physiotherapy and speech therapy

INTERVENTIONS:
Procedure: Physiotherapy and speech therapy

SUMMARY:
This is a prospective study of patients with stroke with accompanying motor and visual deficits. There will be patients' evaluations at 2 time points at the acute and subacute period after the stroke. Statistical correlation of the improvement of their deficits will be conducted

ELIGIBILITY:
Inclusion Criteria:

acute phase stroke patients with motor and visual deficits

Exclusion Criteria:

previous stroke, neurologic disease or visual deficit

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
hemispheric stroke scale | participants will be followed for the duration of hospital stay, an expected average of 6 weeks from the time of stroke
visual fields exam | participants will be followed for the duration of hospital stay, an expected average of 6 weeks from the time of stroke

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece